CLINICAL TRIAL: NCT05765591
Title: Effects of Balneotherapy for Patients With Post-COVID Syndrome
Brief Title: Balneotherapy for Patients With Post-acute Coronavirus Disease (COVID) Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Caldes de Montbui's City Council (Unknown); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Xavier Nogués Solan, Translational Clinical Research Program Coordinator, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/10072/I
Record Dates: First submitted 2023-03-09; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Post-COVID-19 Syndrome
Keywords: Balneotherapy; Post-COVID-19 syndrome; Patient Reported Outcome Measures
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Balneology

STUDY DESIGN:
Intervention Model Description: Randomized controlled longitudinal interventional study
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balneotherapy group (Experimental): The patients allocated to the Balneotherapy group were subject to 3 weekly sessions of Balneotherapy together with an structured program of aquatic exercises on alternate days in groups of 8 during 4 weeks. The weekly planning was structured as following:
  1. st day: Pool, shower, inhalation and aquatic exercises
  2. nd day: Pool, shower, inhalation.
  3. rd day: Pool, shower, inhalation and aquatic exercises
  Interventions: Other: Balneotherapy and aquatic exercises
- Control group (No Intervention): Patients from the control group were instructed to not participate in any BT-related activity during the duration of the study and to continue with usual care and activities

INTERVENTIONS:
Other: Balneotherapy and aquatic exercises — Information has already been included in arm/group descriptions
  Arms: Balneotherapy group

SUMMARY:
The goal of this randomized controlled study is to evaluate the effects of balneotherapy (BT) and aquatic exercises in patients with post-acute COVID syndrome (PACS). The main question it aims to answer are:

• Does BT and aquatic exercises alleviate some of the most prevalent features that characterize post-acute COVID syndrome?

Participants allocated to the intervention group will undergo 3 weekly sessions of BT and aquatic exercises on alternate days in groups of 8 during 4 weeks. Prior the beginning of the intervention, patients were asked to complete an array of validated self-reported questionnaires that covered an important part of PACS symptomatology. These patients were asked to complete these same questionnaires immediately after completing the intervention and one month after. They were also asked to report adverse events associated to the intervention.

Patients allocated to the control group were asked to complete the same questionnaires at baseline and one and two months post-baseline. They were instructed to not enroll in any kind of BT-related activities during the duration of the study.

Questionnaires were analyzed and compared between groups to assess the effects of the intervention.

DETAILED DESCRIPTION:
Participants were recruited in the multidisciplinary Post-COVID unit of the Hospital del Mar or in a primary care center in Barcelona (Spain). In addition, Caldes de Montbui's City Council also advertised the project for patient recruitment on its public website. Inclusion criteria were individuals ≥18 years old with a PACS diagnosis provided by a physician.

Exclusion criteria included patients with preexisting disorders to the severe acute respiratory syndrome (SARS) coronavirus (CoV) 2 infection that displayed an important clinical overlap with PACS i.e., fibromyalgia (FM), chronic fatigue syndrome, chronic pain, and generalized anxiety disorder and/or depression that required pharmacological treatment. Patients with chronic debilitating conditions that required active treatment were also excluded i.e. cancer, chronic viral infections, systemic autoimmune diseases, epilepsy, uncontrolled endocrine disorders, etc. Patients with fear of water, incontinence, severe venous insufficiency, physical disabilities that hindered performance of Balneotherapy (BT)/aquatic exercises, and those who reported a tendency for symptomatic low blood pressure were also excluded. Blood tests performed within 4 months or less before the initial visit were mandatory for preselection and were reviewed: patients with anaemia, chronic kidney disease (CKD) stage 4 or less, chronic liver insufficiency, thyroid function abnormalities, and in general, any significant blood test abnormality that could be associated with PACS-related symptomatology were excluded.

Included patients underwent initial visit in which clinical data was reviewed and registered. Participants were randomly assigned to the intervention or control group through a lottery method. Patients were asked to not vary their usual care or initiate any other kind of therapy during the duration of the study. Post-Acute COVID symptoms At the time of the initial visit several clinical parameters were registered including: age, sex Body Mass Index (BMI), date of SARS-CoV-2 infection, admission into the Intensive Care Unit (yes/no), Visual Analogue Scale (VAS), and a large array of PACS-related symptoms(yes/no) that were classified according to the system/organ affected

Study design The study was designed as a prospective randomized controlled study. Data was collected at 3 time points: 1) initial visit (baseline), 2) at the end of BT or one month after baseline in control group, and 3) one month after BT finalization or two months after baseline in control group. Balneotherapy (BT) intervention The BT intervention consisted of 3 weekly sessions on alternate days in groups of 8 during 4 weeks, i.e., 12 sessions in total. The weekly planning was structured as following:

1 st day: Pool, shower, inhalation and aquatic exercise 2 nd day: Pool, shower, inhalation. 3 rd day: Pool, shower, inhalation and aquatic exercise The exercise program was designed by qualified specialists from the Caldes de Montbui spa. Exercises were performed in the thermal water pool, at 32°C during 2 hours. At the start of the session, patients were instructed to inhale thermal water vapor for 10 minutes, alternating between nose and mouth. Subsequently they underwent a circular shower during 10 minutes with a very fine jet that ran from the ankles to the neck to activate circulation. The temperature of the water and the power of the jet was set by the patient.

Next, they started the exercise program which lasted 15 minutes and was structured as follows:

1. Ankle joints workout, knee flexions, and abductors workout.
2. Waist and arm rotation.
3. Arm raise exercises: arms were raised and lowered from legs to mid-waist. Subsequently, the same exercise was repeated but raising concomitantly knees and, if possible, clapping hands above the head.
4. Hand exercises: patients were instructed to open and close their hands first, and then, repeated the same exercise but alternating hiding or exposing their thumbs.
5. Lateral neck movements.
6. Cycling and rowing movements while holding onto the pool's wall.
7. Walking 2 laps around the pool. During the last 15-20 minutes patients were allowed to relax in the whirlpool.

Control group Patients from the control group were instructed to not participate in any BT-related activity during the duration of the study and to continue with usual care and activities.

Primary Outcome To evaluate the effects of BT we employed an array of validated self-reported questionnaires that covered an important part of PACS symptomatology. The primary outcome of the study was to evaluate differences in questionnaire scores from baseline between both groups. The following scales and questionnaires were employed:

1. Post-COVID-19 functional status scale (PCFS)
2. Modified Medical Research Council (mMRC) Dyspnoea Scale
3. Short Form-36 Health Survey (SF-36) to evaluate generic health-related quality of life (HRQL)
4. Pittsburgh Sleep Quality Index (PSQI)
5. Hospital Anxiety and Depression Scale (HADS)
6. Memory failures in everyday life following severe head injury (MFE-30)
7. Visual Analogic Scale (VAS) Secondary outcomes The percentage of individuals within each group that showed any improvement in the questionnaires' scores at timepoints 2 and 3 compared to baseline were also calculated and compared between groups.

Statistical methods Descriptive statistics were used for demographic and clinical characteristics related to PACS. Comparisons between groups for quantitative variables were performed by t-test and chi-square tests were used for qualitative variables. Questionnaire scores were analysed using the intra-individual absolute change between baseline and post-BT or one month after baseline (control group), and between baseline and one month after completing BT or two months after baseline (control group). One-way ANOVA or chi-square were used for comparisons between groups. The change between time points was also categorized according to whether score improvement was observed (yes/no).

Chi-square test was used to perform the corresponding comparisons between groups.

Finally, univariate General Linear Model (GLM) or multinomial logistic regression were used for group comparisons adjusted by age and BMI. Statistical analysis was done with Statistical Package for the Social Sciences (SPSS) Statistics version 22.0. P values lower than 0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥18 years old with a post-acute COVID-19 syndrome diagnosis provided by a physician.

Exclusion Criteria:

* Patients with preexisting disorders to the acute SARS-CoV-2 infection that displayed an important clinical overlap with PACS i.e., fibromyalgia (FM), chronic fatigue syndrome, chronic pain, and generalized anxiety disorder and/or depression that required pharmacological treatment. Patients with chronic debilitating conditions that required active treatment were also excluded i.e. cancer, chronic viral infections, systemic autoimmune diseases, epilepsy, uncontrolled endocrine disorders, etc. Patients with fear of water, incontinence, severe venous insufficiency, physical disabilities that hindered performance of balneotherapy/aquatic exercises, and those who reported a tendency for symptomatic low blood pressure were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Differences in questionnaire scores in follow-up time points compared to baseline between both groups | 2 months i.e., baseline, post-balneotherapy (or one month post-baseline in the control group), and 1 month post-balneotherapy (or 2 months post-baseline in the control group)
  To evaluate the effects of BT we employed an array of validated self-reported questionnaires that covered an important part of PACS symptomatology. The primary outcome of the study was to evaluate differences in questionnaire scores from baseline between both groups. The following scales and questionnaires were employed:
  1. Post-COVID-19 functional status scale (PCFS)
  2. mMRC (Modified Medical Research Council) Dyspnoea Scale
  3. Short Form-36 Health Survey (SF-36)
  4. Pittsburgh Sleep Quality Index (PSQI)
  5. Hospital Anxiety and Depression Scale (HADS)
  6. Memory failures in everyday life following severe head injury (MFE-30)
  7. Visual Analogic Scale (VAS)

SECONDARY OUTCOMES:
Differences in the percentage of individuals within each group that showed any improvement in the questionnaires' scores at follow-up time-points compared to baseline | 2 months i.e., baseline, post-balneotherapy (or one month post-baseline in the control group), and 1 month post-balneotherapy (or 2 months post-baseline in the control group)
  Differences in the percentage of individuals within each group that showed any improvement in the questionnaires' scores at follow-up time-points compared to baseline. The following scales and questionnaires were employed:
  1. Post-COVID-19 functional status scale (PCFS)
  2. mMRC (Modified Medical Research Council) Dyspnoea Scale
  3. Short Form-36 Health Survey (SF-36)
  4. Pittsburgh Sleep Quality Index (PSQI)
  5. Hospital Anxiety and Depression Scale (HADS)
  6. Memory failures in everyday life following severe head injury (MFE-30)
  7. Visual Analogic Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar Medical Research Institute, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
This is a closed study and there is no plan to share individual participant data.

REFERENCES:
- [Derived] Ovejero D, Ribes A, Villar-Garcia J, Trenchs-Rodriguez M, Lopez D, Nogues X, Guerri-Fernandez R, Garcia-Giralt N. Balneotherapy for the treatment of post-COVID syndrome: a randomized controlled trial. BMC Complement Med Ther. 2025 Feb 4;25(1):37. doi: 10.1186/s12906-025-04784-3. PMID 39905419